CLINICAL TRIAL: NCT00238446
Title: A Prospective, Open-label, Multicenter Extension Study on the Efficacy and Safety of Enteric-coated Mycophenolate Sodium (EC-MPS) in Heart Transplant Recipients
Brief Title: Efficacy and Safety of Enteric-coated Mycophenolate Sodium in Heart Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CERL080A2401E1
Record Dates: First submitted 2005-10-11; First posted 2005-10-13 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Patients Successfully Completing the 12-month Treatment Period of the Core Study (de Novo Heart Recipients) Who Were Interested of Being Treated With EC-MPS
Keywords: Enteric-coated mycophenolate sodium, heart transplant recipients, long term safety

INTERVENTIONS:
Drug: EC-MPS

SUMMARY:
This purpose of this extension study of patients being treated with EC-MPS is to assess the long term safety of this medication.

ELIGIBILITY:
Inclusion Criteria:

Patients who were participating in the core study CERL080A2401 and have successfully completed the first 12 months of the core study

Exclusion Criteria:

Patients who did not complete the 12-month core study CERL080A2401

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2003-04; Primary Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis